CLINICAL TRIAL: NCT01786473
Title: A Multi-center, Double Blind, Randomized, Placebo Controlled Study of Testogel® (Testosterone Gel 50mg/5g) in the Treatment of Male Hypogonadism
Brief Title: Testogel® (Testosterone Gel 50mg/5g) in the Treatment of Male Hypogonadism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires Besins International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01BHR11
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testogel 1% 5g QD (Experimental)
  Interventions: Drug: Testogel 1%
- Placebo gel 5g QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testogel 1%
  Arms: Testogel 1% 5g QD
Drug: Placebo
  Arms: Placebo gel 5g QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Testogel® 50mg/5g gel administered once daily (QD, morning dosing) compared to placebo administered once daily (QD, morning dosing), for 3 months, in hypogonadal men with testosterone deficiency being confirmed by clinical features and biochemical tests. For men with hypogonadism, treatment aims to restore testosterone levels to normal physiological range.

ELIGIBILITY:
Inclusion Criteria:

* Male ages 18-68 years diagnosed as having testosterone deficiency with clinical symptoms
* A morning (8:00-10:00) serum Total Testosterone concentration of ≤ 300 ng/dL, confirmed by a second measurement of morning serum Total Testosterone concentration ≤ 300 ng/dL (samples to be taken 1 - 3 weeks apart)

Exclusion Criteria:

* Abnormal prostate as evidenced by prostatic symptoms, prostatic masses or induration on rectal examination, or elevated levels of prostate specific antigen (PSA > 4ng/ml) or a maximum urine flow rate of less than 12 ml/sec(of a urine volume greater than 150ml) (and/or an International Prostate Symptom Score IPSS score >19)
* Hematocrit > 50%
* Major psychiatric illness
* Unable to understand the protocol or to give informed consent
* Use of paroxetine and clomipramine
* Active alcoholism
* History of drug abuse within the past five years;
* Use of drugs that might interfere with the results of the study (e.g., antiandrogen, estrogens or P 450 enzyme inducers, barbiturates);
* BMI < 18 or > 30 according to Chinese BMI references;
* Generalized skin disease that may affect absorption of T (e.g., psoriasis) or a known skin intolerance to alcohol;
* Prolactin > 40 mcg/L;
* Untreated severe obstructive sleep apnea;.
* Uncontrolled or poorly controlled heart failure

Ages: 18 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with morning serum Total Testosterone concentration within the physiological range (300 - 1000 ng/dL or 10.4 - 34.7 nmol/L) after 3 months of Testogel treatment compared to placebo-treatment | 3 months

SECONDARY OUTCOMES:
morning serum Total Testosterone (TT) concentration compared to placebo treatment | 3 months
morning serum Total Testosterone (TT) concentration compared to baseline values | 3 months
serum concentrations of TT, calculated free testosterone (cFT), DHT, E2, LH, and FSH, SHBG | 3 months
prostate assessments (PSA, urine flow rate, DRE, ultrasound B) | 3 months
skin integrity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China